CLINICAL TRIAL: NCT06566378
Title: The Effect of Cold Application and Vibration in Reducing Pain During Vaccination in Children: A Randomized Controlled Study
Brief Title: Effect of Cold Application and Vibration in Reducing Pain During Vaccination in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO 2024/175
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pain; Pain, Acute; Vaccination; Children; Cold Application; Vibration
Keywords: pain; Vaccination; Child; Cold Application; Vibration; Buzzy
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Intervention Model Description: This prospective, randomised controlled study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placed under arm Buzzy Group (Experimental): In children pre-procedure, buzzy was placed under the armpit. The children were made before starting the application. It continued until the end of vaccination procedure.
  Interventions: Device: Buzzy
- Placed in standard Buzzy Group (Experimental): In children pre-procedure, buzzy was placed on the arm. The children were made before starting the application. It continued until the end of vaccination procedure.
  Interventions: Device: Buzzy (Placed in standard)
- Control Group (No Intervention): In this group, children received routine vaccination procedure.

INTERVENTIONS:
Device: Buzzy — In children pre-procedure, buzzy was placed under the armpit. The children were made before starting the application. It continued until the end of vaccination procedure.
  Arms: Placed under arm Buzzy Group
Device: Buzzy (Placed in standard) — In children pre-procedure, buzzy was placed on the arm. The children were made before starting the application. It continued until the end of vaccination procedure.
  Arms: Placed in standard Buzzy Group

SUMMARY:
The study was designed as a randomized controlled experimental research with the purpose of determining the effect of using Cold Application and Vibration in reducing pain during routine vaccination in children.

DETAILED DESCRIPTION:
In the literature, it is stated that nurses should use pharmacological and non-pharmacological methods in pain and anxiety management in painful procedures. Evidence-based studies are needed to show the effectiveness of non-pharmacological methods in reducing pain during invasive procedures and to investigate the effects of easy-to-apply methods on pain.In light of this information, this study aimed to examine the effect of by using Cold Application and Vibration in reducing pain during routine vaccination in children. Cold Application and Vibration will be done with BUZZY.

This study is a prospective, randomized and controlled trial. Children aged 13 years who required routine vaccination were divided into three groups; placed under arm Buzzy, placed in standard Buzzy, and Control. Data were obtained through face-to-face interviews with the children, their parents, and the observer before and after the procedure. The children's pain levels were assessed and reported by the parents and observers and the children themselves who selfreported using Wong-Baker FACES.

The study population consisted of the children's during routine vaccination in children aged 13 years. Sample of the study consisted of a total of 90 children who met the sample selection criteria and were selected via randomization method.

Children were randomized into three groups; placed under arm Buzzy (n:30), placed in standard Buzzy (n:30), and Control (n:30). Data were collected using the Interview and Observation Form and Wong-Baker FACES Pain Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Children the ages of 13 years (planned to be included in the vaccination calendar program),
* Volunteering of the child and parent to participate in the study,
* Healthy children,
* Vaccination should be done by the same nurse,

Exclusion Criteria:

* The child has any acute or chronic disease,
* The child has a mental disability, vision, speech or communication problems,
* The parent has hearing, vision or verbal communication difficulties,
* The child used analgesics in the last 6 hours,
* Infection, disruption of skin integrity and rash in the area where theapplication will be made,
* Exclusion criteria were that the parent or child wanted to leave the study at any point.

Ages: 13 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | Through study completion, an average of 1 year
  In the study, pain level evaluations, the children's self-evaluations, parents' evaluations and the researcher's evaluations were carried out using the WB-FACES scale. This scale was developed by Donna Wong and Connie Morain Baker in 1988. The scale is graded between 0-10 points. A smiling face on the far left symbolizes "no pain" (0 very happy/no pain) and the pain increases from left to right. On the other hand, a crying face on the far right symbolizes "unbearable pain" (10 'hurts worst'). As the numbers increase in this scoring system, facial expressions also change referring to an increase in pain levels.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, PhD., Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Bucak, Burdur, Bucak, Turkey (Türkiye)

REFERENCES:
- [Derived] Ates Besirik S, Turgut MA, Sahiner NC, Baxter AL, Kirboga Z. Reducing vaccination pain using a multidermatomal or deltoid region buzzy(R) applications versus control: A randomized controlled study. J Pediatr Nurs. 2025 Nov-Dec;85:783-791. doi: 10.1016/j.pedn.2025.10.011. Epub 2025 Oct 27. PMID 41151224